CLINICAL TRIAL: NCT03026140
Title: Neoadjuvant Immune Checkpoint Inhibition and Novel IO Combinations in Early-stage Colon Cancer (Amended Protocol of: Nivolumab, Ipilimumab and COX2-inhibition in Early Stage Colon Cancer: an Unbiased Approach for Signals of Sensitivity: The NICHE TRIAL)
Brief Title: Neoadjuvant Immune Checkpoint Inhibition and Novel IO Combinations in Early-stage Colon Cancer
Acronym: NICHE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N16NCI; 2024-513314-35-00 (EU CTIS Number)
Record Dates: First submitted 2016-12-15; First posted 2017-01-20 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-06

CONDITIONS: Colon Carcinoma
Keywords: MSI tumors; MSS tumors; short-term immunotherapy; surgical resection; nivolumab; ipilimumab; COX2; Anti-IL8; Relatlimab; Anti-LAG3
MeSH Terms: conditions — Colonic Neoplasms | interventions — Nivolumab; Ipilimumab; Celecoxib; HuMax-IL8; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- group 1 - closed (Experimental): drug: ipilimumab 1 mg/kg day 1 (IV) drug: nivolumab 3 mg/kg on day 1 and day 15 (IV)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- group 2 - closed (Experimental): drug: ipilimumab 1 mg/kg day 1 (IV) drug: nivolumab 3 mg/kg on day 1 and day 15 (IV) drug: celecoxib 200 mg daily (oral)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Celecoxib 200mg
- Anti-IL8 cohort 4 (pMMR/MSS tumors) - closed (Experimental): drug: nivolumab 3 mg/kg day 1 and day 15 (IV) drug: BMS-986253 (anti-IL8) 2400mg on day 1 and day 15 (IV)
  Interventions: Drug: Nivolumab; Drug: BMS-986253
- Relatlimab cohort 5 (pMMR/MSS tumors) (Experimental): drug: nivolumab 240mg IV on day 1 and day 15 drug: relatlimab 240mg IV on day 1 and day 15
  Interventions: Drug: Nivolumab; Drug: BMS-986016
- Relatlimab cohort 6 (dMMR/MSI tumors) - closed (Experimental): drug: nivolumab 480mg IV on day 1 and day 29 drug: relatlimab 480mg IV on day 1 and day 29
  Interventions: Drug: Nivolumab; Drug: BMS-986016
- Cohort 7 - dMMR - 3 cycles neoadjuvant nivolumab + relatlimab (Experimental): Patients with dMMR tumors will be treated with 3 cycles of neoadjuvant nivolumab (480mg) + relatlimab (160mg) on day 1, day 29 and day 57 followed by surgery within 12 weeks and not earlier than 10 weeks from enrollment
  Interventions: Drug: Nivolumab; Drug: BMS-986016
- Cohort 8 - dMMR - 3 cycles neoadjuvant nivolumab (Experimental): Patients with dMMR tumors will be treated with 3 cycles of neoadjuvant nivolumab (480mg) on day 1, day 29 and day 57 followed by surgery within 12 weeks and not earlier than 10 weeks from enrollment.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3mg/kg (day 1 and day 15), administered neoadjuvant before surgery
  Other Names: nivolumab (opdivo)
Drug: Ipilimumab — Ipilimumab 1 mg/kg (day 1) ,administered neoadjuvant before surgery
  Other Names: Ipilimumab (Yervoy)
  Arms: group 1 - closed; group 2 - closed
Drug: Celecoxib 200mg — celecoxib will be administered starting day 1 until 1 day before surgery daily (if patient is randomized to group 2 (only applicable for patients with a MSS tumor)
  Other Names: Celebrex
  Arms: group 2 - closed
Drug: BMS-986253 — BMS-986253 2400mg IV will be administered on day 1 and 15 (only applicable for patients with MSS tumors)
  Other Names: Anti-IL8
  Arms: Anti-IL8 cohort 4 (pMMR/MSS tumors) - closed
Drug: BMS-986016 — Relatlimab will be administered IV, in cohort 5 240mg on day 1 and day 15, in cohort 6 480mg on day 1 and day 29, in cohort 7 160mg on day 1, day 29 and day 57
  Other Names: Relatlimab
  Arms: Cohort 7 - dMMR - 3 cycles neoadjuvant nivolumab + relatlimab; Relatlimab cohort 5 (pMMR/MSS tumors); Relatlimab cohort 6 (dMMR/MSI tumors) - closed

SUMMARY:
In this exploratory study, patients with stage 1-3 adenocarcinoma of the colon with no signs of distant metastases will be treated with short-term immunotherapy + novel IO combinations (i.e. anti-IL 8, COX2-inhibitors, anti-LAG3). This treatment will be given during the window period until surgical resection of the tumor. The duration of treatment will be in between approximately 6 and 12 weeks.

DETAILED DESCRIPTION:
In this multi-center, open-label, exploratory study, the investigators will enroll 60 patients within two years, including 30 patients with MSS tumors and 30 patients with MSI tumors. Patients with MSS tumors will be randomized to either group 1 or 2. Patients with MSI tumors will all be allocated to group 1.

Patients in group 1 will be treated with a single dose of ipilimumab 1mg/kg on day 1 and two cycles of nivolumab 3mg/kg on day 1 and 15, respectively.

Patients in group 2 will be treated with a single dose of ipilimumab 1mg/kg on day 1, two cycles of nivolumab 3mg/kg one day 1 and 15 and celecoxib daily until the day before surgery.

The study was amended in May 2020 to enroll an additional 70 patients in the MSI cohort after the first 30 patients, making a total of 100 patients with MSI tumors. A formal sample size calculation and primary endpoint of 3-year disease-free-survival (DFS) for this group was added.

The study was amended in July 2021 to add a new cohort, cohort 4, for patients with pMMR/MSS tumors. Once accrual of 30 evaluable patients in group 2 was completed, a new cohort opened in which patients will receive nivolumab plus anti-IL8 (BMS-986253).

The study was amended in November 2022 to add cohort 5 and 6, both in which patients will receive nivolumab plus relatlimab (anti-LAG3). Patients with pMMR/MSS tumors will be randomized 1:1 between cohort 4 and cohort 5, patients with dMMR/MSI tumors will be enrolled in cohort 6.

Accrual for cohort 4 was reached in July 2023. In April 2024, accrual for cohort 6 was reached. Per April 2024 only cohort 5 is open for recruitment.

The study was amended in April 2025 to add cohort 7 and 8. Patients with dMMR/MSI tumors will be randomized 1:1 between cohort 7 and 8, in which they will receive 3 cycles of nivolumab + relatlimab or 3 cycles of nivolumab monotherapy respectively. Per June 2025, cohort 5, 7 and 8 are open for recruitment.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent
* Patients at least 18 years of age
* Non-metastatic adenocarcinoma of the colon (and rectosigmoid considered as nonrectal and not undergoing neoadjuvant treatment)

  * No signs of distant metastases on CT-scan and physical examination;
  * dMMR cohorts 3+6: >cT3 and/or N+

Exclusion criteria:

* No signs of distant metastases
* No signs of obstruction or macroscopic bleeding or suspicion of perforation
* Colonoscopy must be performed after registration to obtain study-specific biopsies. If biopsies are not possible, patients cannot be included in the study
* WHO performance status of 0 or 1
* No previous treatment with immune checkpoint inhibitors targeting CTLA-4, PD-1 or PD-L1
* For patients with MSS tumors: no current use of NSAIDs or COX2-inhibitors at registration and no active peptic ulcer, gastrointestinal bleeding, unstable ischemic heart disease of thrombus etiology or significant established ischemic heart disease, peripheral arterial disease and/or cerebrovascular disease
* No radiotherapy prior to or planned post-surgery radiotherapy
* No history of allergy to study drug components, severe hypersensitivity reaction to any monoclonal antibody, allergy or severe hypersensitivity to NSAIDs or COX2-I (MSS tumors)
* No intercurrent illnesses, including but not limited to infections, unstable angina pectoris
* No positive test for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* No autoimmune disease
* No conditions requiring systemic treatment with either corticosteroids (10 mg daily prednisone or more and equivalents) or other immunosuppressive medications within 14 days of study drug administration
* No live vaccines in the 4 weeks prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2032-03-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events during the treatment and follow-up (safety) | until 100 days after last patient last study drug treatment
  Adverse events will be assessed (according to CTCAE v4.0) during treatment and follow-up.
Disease free survival | until 5 years after diagnosis
  To assess efficacy of neoadjuvant ipilimumab plus nivolumab in terms of disease-free survival
Major Pathological Response | From date of randomization until the date of first documented progression, assessed up to 63 months
  To assess efficacy of neoadjuvant nivolumab monotherapy and neoadjuvant nivolumab plus relatlimab in terms of major pathologic response

SECONDARY OUTCOMES:
Immune activating capacity of short-term pre-operative immunotherapy | within 2 years after study completion
  identify underlying potential escape mechanisms by comparing pre-treatment and post-treatment biopsies
Relapse free survival | 3-5 years after last patient inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Chalabi, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (6):
- Netherlands (6):
  - Marieke van de Belt, Amsterdam
  - OLVG, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Spaarne Ziekenhuis, Haarlem
  - Tergooi, Hilversum
  - Haga ziekenhuis, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan PB, Verschoor YL, van den Berg JG, Balduzzi S, Kok NFM, Ijsselsteijn ME, Moore K, Jurdi A, Tin A, Kaptein P, van Leerdam ME, Haanen JBAG, Voest EE, de Miranda NFCC, Schumacher TN, Wessels LFA, Chalabi M. Neoadjuvant immunotherapy in mismatch-repair-proficient colon cancers. Nature. 2025 Dec;648(8094):726-735. doi: 10.1038/s41586-025-09679-4. Epub 2025 Oct 20. PMID 41115454
- [Derived] de Gooyer PGM, Verschoor YL, van den Dungen LDW, Balduzzi S, Marsman HA, Geukes Foppen MH, Grootscholten C, Dokter S, den Hartog AG, Verbeek WHM, Woensdregt K, van den Broek JJ, Oosterling SJ, Schumacher TN, Kuhlmann KFD, Beets-Tan RGH, Haanen JBAG, van Leerdam ME, van den Berg JG, Chalabi M. Neoadjuvant nivolumab and relatlimab in locally advanced MMR-deficient colon cancer: a phase 2 trial. Nat Med. 2024 Nov;30(11):3284-3290. doi: 10.1038/s41591-024-03250-w. Epub 2024 Sep 15. PMID 39278994
- [Derived] Cercek A. Neoadjuvant Treatment of Mismatch Repair-Deficient Colon Cancer - Clinically Meaningful? N Engl J Med. 2024 Jun 6;390(21):2024-2025. doi: 10.1056/NEJMe2404601. No abstract available. PMID 38838316
- [Derived] Chalabi M, Verschoor YL, Tan PB, Balduzzi S, Van Lent AU, Grootscholten C, Dokter S, Buller NV, Grotenhuis BA, Kuhlmann K, Burger JW, Huibregtse IL, Aukema TS, Hendriks ER, Oosterling SJ, Snaebjornsson P, Voest EE, Wessels LF, Beets-Tan RG, Van Leerdam ME, Schumacher TN, van den Berg JG, Beets GL, Haanen JB. Neoadjuvant Immunotherapy in Locally Advanced Mismatch Repair-Deficient Colon Cancer. N Engl J Med. 2024 Jun 6;390(21):1949-1958. doi: 10.1056/NEJMoa2400634. PMID 38838311
- [Derived] Wang D, Cabalag CS, Clemons NJ, DuBois RN. Cyclooxygenases and Prostaglandins in Tumor Immunology and Microenvironment of Gastrointestinal Cancer. Gastroenterology. 2021 Dec;161(6):1813-1829. doi: 10.1053/j.gastro.2021.09.059. Epub 2021 Oct 2. PMID 34606846
- [Derived] Chalabi M, Fanchi LF, Dijkstra KK, Van den Berg JG, Aalbers AG, Sikorska K, Lopez-Yurda M, Grootscholten C, Beets GL, Snaebjornsson P, Maas M, Mertz M, Veninga V, Bounova G, Broeks A, Beets-Tan RG, de Wijkerslooth TR, van Lent AU, Marsman HA, Nuijten E, Kok NF, Kuiper M, Verbeek WH, Kok M, Van Leerdam ME, Schumacher TN, Voest EE, Haanen JB. Neoadjuvant immunotherapy leads to pathological responses in MMR-proficient and MMR-deficient early-stage colon cancers. Nat Med. 2020 Apr;26(4):566-576. doi: 10.1038/s41591-020-0805-8. Epub 2020 Apr 6. PMID 32251400